CLINICAL TRIAL: NCT06397807
Title: Postoperative Pain Management on Patients Undergoing Video-assisted Thoracoscopic (VATS) Lung Tumor Resection: a Prospective Cohort Study
Brief Title: Postoperative Pain Management on Patients Undergoing Lung Tumor Resection
Status: Not yet recruiting | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hsin-Yuan Fang, Associate Director of China Medical University Hospital, China Medical University Hospital
Other Study IDs: CMUH-112-01
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain; Lung Cancer; Lung Tumor
Keywords: Video-assisted thoracoscopic (VATS) lung tumor resection; Naldebain; Dinalbuphine sebacate; Multimodal analgesia; Enhanced Recovery After Surgery; ERAS; MMA
MeSH Terms: conditions — Pain, Postoperative; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NALDEBAIN: Patients injected with dinalbuphine sebacate intramuscularly will be allocated to NALDEBAIN group.
  Interventions: Drug: Dinalbuphine sebacate; Drug: Analgesic injectables; Drug: Enteral analgesics
- CONTROL: Patients receiving postoperative pain management without dinalbuphine sebacate will be allocated to CONTROL group.
  Interventions: Drug: Analgesic injectables; Drug: Enteral analgesics

INTERVENTIONS:
Drug: Dinalbuphine sebacate — Dinalbuphine sebacate (DS) is a long-acting injectable. With oil-based formulation, DS will slowly releases to blood vessel and be hydrolyzed to nalbuphine after intramuscularly injection. The analgesic effect lasts around 5 to 7 days.
  Other Names: Naldebain
  Groups: NALDEBAIN
Drug: Analgesic injectables — Opioids, NSAIDs or acetamol will be administrated as need.
  Other Names: A.I.
Drug: Enteral analgesics — Opioids, NSAIDs or acetaminophen will be prescribed if necessary.
  Other Names: E.A.

SUMMARY:
Multimodal analgesia (MMA) is an essential part of Enhanced Recovery After Surgery (ERAS) protocol. The principle of MMA is to manage pain with analgesics of multiple classes acting on distinct target sites through different strategies. MMA can reduce the adverse reaction caused by opioids and improve the quality of recovery from surgery. Inadequate postoperative pain management will increase the risk of complications, including pneumonia, deep vein thrombosis, infection, delayed surgical healing, and chronic postoperative pain.

DETAILED DESCRIPTION:
This prospective, observational study is planned to investigate the efficacy of different MMA regimens conducting in our hospital. Patients undergoing video-assisted thoracoscopic (VATS) lung tumor resection will be invited to participate in the study and grouped based on the MMA regimens. Anxiety, quality of recovery, pain intensity will be evaluated pre- and post-operatively. Demographic data, surgery record, medicine record and postoperative complications will be gained from medical history system and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. aged above 18.
2. diagnosed as lung cancer.
3. planning to undergo primary, video-assisted thoracoscopic lung tumor resection.
4. American Society of Anesthesiology Physical Class 1~3.

Exclusion Criteria:

1. unable to take assessments of the endpoints.
2. having this surgery in an emergency.
3. surgery involving other orangs, such as esophagus and stomach.
4. severe abnormality of cardiac, hepatic, or renal function.
5. allergic to opioids.
6. allergic to NSAIDs.
7. diagnosed as chronic pain or chronic use of analgesics.
8. unsuitable for participation judged by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient scheduled to have video-assisted thoracoscopic lung tumor resection in China Medical University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | Within 3 days after surgery
  Pain intensity is assessed by numerical rating scale (NRS) daily during hospital stay after delivery. NRS is a 11-point scale which labeled from zero (no pain) to ten (worst pain). The area under the curve of NRS are calculated.

SECONDARY OUTCOMES:
Consumption of analgesics | Within 7 days after surgery
  The mean total consumption of analgesics during the hospital stay after delivery.
GAD-7 | At baseline, 7 days and 3 months after surgery
  This self-administered patient questionnaire is used as a screening tool and severity measure for generalised anxiety disorder (GAD). Respondents are asked to rate each item for frequency of occurrence using a 4-point Likert scale (Not at all = 0, Several days = 1, More than half the days = 2, and Nearly every day = 3). All responses are summed to calculate the total GAD-7 score.
QoR-15 | At baseline, 7 days and 3 months after surgery
  The quality of recovery-15 (QoR-15) is a patient-reported outcome measurement measuring QoR after surgery and anesthesia. The scale is arbitrary and ranges from 0 (extremely poor QoR) to 150 (excellent QoR).

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Yuan Fang, Principal Investigator — China Medical University Hospital; Po-Han Li, Principal Investigator — China Medical University Hospital; Kin-Shing Poon, Principal Investigator — China Medical University Hospital; Hsiurong Liao, Principal Investigator — China Medical University Hospital; Tzu-Min Huang, Principal Investigator — China Medical University Hospital; Yu-Cheng Shen, Principal Investigator — China Medical University Hospital